CLINICAL TRIAL: NCT05555784
Title: Evaluation of Impact of Disease and Visual Disability on Quality of Life and Loss of Independence of Patients Living in France With Leber's Hereditary Optic Neuropathy (LHON) Through Qualitative and Quantitative Data Collection
Status: Completed | Type: Observational
Sponsor: Argo Sante (Other)
Collaborators: GenSight Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A00552-41
Record Dates: First submitted 2022-09-02; First posted 2022-09-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Leber's Hereditary Optic Neuropathy (LHON)
Keywords: Leber's hereditary optic neuropathy (LHON), quality of life, loss of independence, social life, family, socio-professional, France
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Leber's hereditary optic neuropathy (LHON) is a rare mitochondrial genetic disorder characterized by optic nerve atrophy due to the degeneration of retinal ganglion cells, which leads to acute visual loss.

Males are more likely to develop optic neuropathy than women. They experience blurring or clouding of vision in one eye. The fellow eye develops similar symptoms sequentially with a delay of weeks.

This sudden vision loss has devastating consequences on the life course of young men, with the impact of LHON on their quality of life and loss of independence.

Yet, data describing the impacts of LHON on the life-course of patients is lacking, with very little data available in the literature.

This study aims to understand the life of patients living with LHON disease through the analysis of the impact of LHON on the quality of life and loss of independence of patients living in France and to accurately describe the consequences of the disease on their social, familial and professional life.

DETAILED DESCRIPTION:
The protocol presents a retrospective study. Patients living in France with LOHN shall be informed about it and offered to enroll through patients' associations or experts involved. As part of the consent process, participants should be informed of the nature of the study and the objectives and that the replies would remain confidential and anonymous.

After a brief screening, the study divides into two parts: one aiming at collecting quantitative data through 3 standard quality of life questionnaires, and one survey specially written for this study (sample of 25 patients, duration 2 hours). The second is a qualitative interview to deep dive into their personal, social, familial, and professional life (10 patients, duration is 50 minutes). The study contains the detailed sections:

* Screening
* A survey specially designed for the study
* Quality of life through EQ-5D-5L
* Quality of life through NEI VFQ- 25, specific for patients suffering from glaucoma
* Quality of life through ARAMAV questionnaire specific for visually impaired people
* An in-depth qualitative interview, specially designed to fit the requirements of the study

ELIGIBILITY:
Inclusion Criteria:

* 20 to 59 years old
* Living in France and fluent in French
* Diagnosed with Leber's hereditary optic neuropathy (LHON) for more than twelve months and less than five years
* Suffering from the mutation ND4 (m.11778G>A)
* Willing to participate in the study

Exclusion Criteria:

* Not willing to participate in the study
* Patients treated/cured with gene therapy rAAV2/2-ND4 (GS010, Lumevoq®)
* Patients diagnosed there are more than five years or less than twelve months
* Patients suffering from disabilities not related to LHON
* Person or person having a member of their family working in ophthalmology-related industries or profession, in clinical research or associations of patients, or involved in health governmental agencies
* Person having difficulties reading or speaking French, unable to answer the questions

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults living in France diagnosed with Leber's hereditary optic neuropathy (LHON) for more than twelve months and less than five years
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Describe the disease impact on quality of life through qualitative data of loss of independence of patients suffering from LHON and living in France | Once at enrollment
  Descriptive analysis of answers given to ad-hoc questionnaire and qualitative analysis of interviews

SECONDARY OUTCOMES:
Measure the general quality of life | Once at enrollment
  The 5-level EQ-5D version (EQ-5D-5L) comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. It gives a score where 1 represents the better life that ones can imagine, and 0 stands for death. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Measure the vision-related quality of life | once at enrollment
  NEIVFQ-25 (National Eye Institute Visual Functioning Questionnaire - 25): a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. It generates the vision-related sub-scales: global vision activities, difficulty with near vision activities, difficulty with distance vision activities, limitations in social functioning due to vision, role limitations due to vision, dependency on others due to vision, mental health symptoms due to vision, driving difficulties, limitations with peripheral and color vision, and ocular pain.
Measure the independence and independence-related quality of life | once at enrollment
  o 13-30 ARAMAV: independence scale comprising 9 daily life activities groups (personal care, meals intake and preparation, domestic care, finances, society life, practical life, outside travel. Each is evaluated regarding the level of realization, the help received, and the level of satisfaction. It gives 2 scores: an independence score where 100 represents an independent person and 0 a totally dependent person and a quality of life score where 100 represents the better quality of life and 0 is the worse quality of life.
Measure the cost of visual loss in terms of economic impact | once at enrollment
  ad-hoc questionnaire
Assess the patient's needs in care and social-economic support | once at enrollment
  ad-hoc questionnaire
Explore the relation between health status and employment conditions, education, and economic situation | once at enrollment
  ad-hoc questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marieke Podevin, PhD, Principal Investigator — Argo Sante
Locations (1):
- Argo Sante, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cui S, Jiang H, Peng J, Wang J, Zhang X. Evaluation of Vision-Related Quality of Life in Chinese Patients With Leber Hereditary Optic Neuropathy and the G11778A Mutation. J Neuroophthalmol. 2019 Mar;39(1):56-59. doi: 10.1097/WNO.0000000000000644. PMID 29554000
- [Background] Kirkman MA, Korsten A, Leonhardt M, Dimitriadis K, De Coo IF, Klopstock T, Griffiths PG, Hudson G, Chinnery PF, Yu-Wai-Man P. Quality of life in patients with leber hereditary optic neuropathy. Invest Ophthalmol Vis Sci. 2009 Jul;50(7):3112-5. doi: 10.1167/iovs.08-3166. Epub 2009 Feb 28. PMID 19255150
- [Background] Newman NJ. Hereditary optic neuropathies: from the mitochondria to the optic nerve. Am J Ophthalmol. 2005 Sep;140(3):517-23. doi: 10.1016/j.ajo.2005.03.017. PMID 16083845
- [Background] Newman NJ, Yu-Wai-Man P, Carelli V, Biousse V, Moster ML, Vignal-Clermont C, Sergott RC, Klopstock T, Sadun AA, Girmens JF, La Morgia C, DeBusk AA, Jurkute N, Priglinger C, Karanjia R, Josse C, Salzmann J, Montestruc F, Roux M, Taiel M, Sahel JA. Intravitreal Gene Therapy vs. Natural History in Patients With Leber Hereditary Optic Neuropathy Carrying the m.11778G>A ND4 Mutation: Systematic Review and Indirect Comparison. Front Neurol. 2021 May 24;12:662838. doi: 10.3389/fneur.2021.662838. eCollection 2021. PMID 34108929
- [Background] Yu-Wai-Man P, Turnbull DM, Chinnery PF. Leber hereditary optic neuropathy. J Med Genet. 2002 Mar;39(3):162-9. doi: 10.1136/jmg.39.3.162. PMID 11897814
- See also: LHON's French patients community's website — https://www.ouvrirlesyeux.org/fr/2022/07/25/etude-fardeau-de-la-maladie-nohl/